CLINICAL TRIAL: NCT01812629
Title: Clinical Management of Children With Chronic Diarrhea
Brief Title: Nutritional Management of Children With Chronic Diarrhea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AH72
Record Dates: First submitted 2013-03-14; First posted 2013-03-18 (Estimated); Last update posted 2013-03-18 (Estimated); Status verified 2013-03

CONDITIONS: Growth and Tolerance Infant Study

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Experimental Infant Formula (Experimental): Complete peptide amino acid-based infant formula
  Interventions: Other: Experimental Infant Formula

INTERVENTIONS:
Other: Experimental Infant Formula — Infant formula to be fed ad libitum
  Other Names: EleCare

SUMMARY:
The study objective is to assess the growth, tolerance and efficacy of a complete amino acid-based medical food in children with chronic diarrhea.

ELIGIBILITY:
Inclusion Criteria:

* Less than or equal to 9 months of age at enrollment
* Candidates for an elemental formula
* Chronic diarrhea and diagnosis of one of the following conditions: short-bowel syndrome, eosinophilic gastroenteritis, food allergy, inflammatory bowel disease, pancreatic disease, protein maldigestion, HIV-advanced disease or other underlying GI disease with chronic diarrhea controlled by a semi-elemental or elemental formula
* Parents agree to feed infant with experimental formula for least 50% of total calories during study period

Exclusion Criteria:

- Any non-approved concomitant study

Max Age: 9 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 19 (Actual)
Dates: Start 1997-07; Primary Completion 1999-06 (Actual); Study Completion 1999-06 (Actual)

PRIMARY OUTCOMES:
Physician determined target outcome | Study Day (SD)1-84
  Outcome dependent on individual subject assessment and may include decreased stool number, decreased vomiting, decreased gas, weight gain, increased caloric intake, increased protein intake, increased serum albumin concentration, increased hemoglobin concentration, better acceptance of supplemental formula.

SECONDARY OUTCOMES:
Dietary Assessment | Study day (SD) 2-4, 5-7, 25-27 and 81-83
  Parent completed record of infant dietary intake.
Gastro-Intestinal Tolerance | Study Day (SD) 2-4, 5-7, 25-27, 81-83
  Parent reported record of incidence of regurgitation.
Stool characteristics | Study Day (SD) 2-4, 5-7, 25-27 and 81-83
  Parent completed diary of stool consistency, frequency/volume.
Blood Chemistry | Study Day (SD) 1 and 84
  Hemoglobin, hematocrit, serum albumin, total protein, urea nitrogen, alkaline phosphatase
Anthropometrics | Study Day (SD) 1, 28 and 84
  Weight and length

CONTACTS AND LOCATIONS:
Overall Officials: Marlene Borschel, PhD, RD, Study Chair — Abbott Nutrition
Locations (2):
- United States (2):
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Johns Hopkins Hospital, Baltimore, Maryland

REFERENCES:
- [Derived] Borschel MW, Antonson DL, Murray ND, Oliva-Hemker M, Mattis LE, Kerzner B, Tolia V, Baggs G. Two single group, prospective, baseline-controlled feeding studies in infants and children with chronic diarrhea fed a hypoallergenic free amino acid-based formula. BMC Pediatr. 2014 May 29;14:136. doi: 10.1186/1471-2431-14-136. PMID 24885833